CLINICAL TRIAL: NCT04575740
Title: Phenotyping Mechanistic Pathways for Adverse Health Outcomes in Sleep Apnea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Ali Azarbarzin, Associate Scientist, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PhenOSA; 1R01HL153874 (NIH)
Record Dates: First submitted 2020-09-16; First posted 2020-10-05 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2024-08

CONDITIONS: Sleep Apnea
Keywords: Sleep apnea; Hypoxic burden; Arousal intensity; Post-event tachycardia; Positive airway pressure; Apnea hypopnea index
MeSH Terms: conditions — Sleep Apnea Syndromes

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Positive Airway Pressure Device (Experimental): All participants will receive PAP therapy
  Interventions: Device: PAP

INTERVENTIONS:
Device: PAP — Positive airway pressure to treat sleep apnea

SUMMARY:
Obstructive sleep apnea (OSA) is a highly prevalent disorder with adverse neurocognitive and cardio-metabolic outcomes. Continuous positive airway pressure (CPAP) is the gold standard therapeutic option to treat airway obstructions during sleep and thus, prevent its adverse cardiovascular and neurocognitive outcomes. Previous clinical trials, however, have largely failed to show a consistent impact of CPAP on these health outcomes.

One of the main limitations of these trials may be the inadequate characterization of OSA and its acute physiological consequences. By characterizing OSA based on the "apnea-hypopnea index (AHI)", there is a potential risk of negative results.

In this trial, the investigators intend to tackle this issue, by better characterization of OSA-related physiological consequences during sleep using physiologically driven metrics to capture the burden of OSA-related hypoxemia ("hypoxic burden"), autonomic response ("heart rate burden"), and sleep fragmentation ("arousal burden").

ELIGIBILITY:
Inclusion criteria:

* Adults aged 21-80 years.
* Participants with a previous diagnosis of moderate to severe obstructive sleep will be eligible to enroll and attend the baseline study. Patients with a total apnea-hypopnea index greater than 15 events/hr on the baseline study will be eligible for further participation.

Exclusion criteria:

* Current treatment for obstructive sleep apnea (including CPAP, oral appliances, supplemental oxygen). Patients must be untreated prior to the baseline visit.
* Use of medications that might depress respiration (including opioids, barbiturates, benzodiazepines, and Z drugs, including zolpidem, zopiclone, eszopiclone, and zaleplon).
* Active use of non-prescription opioids (e.g., cocaine, methamphetamine)
* Uncontrolled medical problem or major organ system disease, which, in the opinion of the investigators (PI and Co-Is), would interfere with the evaluation of the subject (e.g., uncontrolled hypertension, unstable coronary heart disease, etc.).
* History of congestive heart failure, renal insufficiency, systemic neurological condition that could affect respiration.
* Sleep disordered breathing or respiratory disorders other than obstructive sleep apnea:

  * central sleep apnea (>50% of respiratory events scored as central),
  * chronic hypoventilation/hypoxemia (awake SaO2 < 92% by oximetry) due to chronic obstructive pulmonary disease or other respiratory conditions.
* Other sleep disorders: periodic limb movements (periodic limb movement arousal index > 10/hr), narcolepsy, or parasomnias.
* Patients unable or unwilling to use CPAP.
* Insomnia or insufficient sleep (self-reported inability to sleep >6 hrs night).
* Pregnancy (women)

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 209 (Actual)
Dates: Start 2020-09-10 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline flow-mediated vasodilation at 12 weeks | 12 weeks
  Flow mediated vasodilation is studied using high resolution ultrasound of the artery.
Change from baseline 24-hour mean systolic blood pressure at 12 weeks | 12 weeks
  Mean systolic blood pressure over a 24-hour period is measured using an ambulatory blood pressure monitor.
Change from baseline Epworth Sleepiness Scale (ESS) at 12 weeks | 12 weeks
  Self-reported sleepiness measured using the Epworth Sleepiness Scale (units on a scale). Values range from 0-24; higher values indicate greater sleepiness.

SECONDARY OUTCOMES:
Change from baseline F2-Isoprostane/Creatinine Ratio at 12 weeks | 12 weeks
  F2-Isoprostane/Creatinine Ratio, a measure of oxidative stress, is calculated from urine sample.
Change from baseline Albumin/Creatinine Ratio at 12 weeks | 12 weeks
  Urinary Albumin/Creatinine Ratio is calculated from urine samples.
Change from baseline Albumin without Creatinine at 12 weeks | 12 weeks
  Urinary Albumin is calculated from urine samples.
Change from baseline Oxidized low-density lipoprotein (LDL) at 12 weeks | 12 weeks
  Oxidized low-density lipoprotein measurements are calculated through fasting phlebotomy.
Change from baseline N-terminal pro b-type natriuretic peptide (NT-proBNP) at 12 weeks | 12 weeks
  N-terminal pro b-type natriuretic peptide (NT-proBNP) measurements are calculated through fasting phlebotomy.
Change from baseline Hemoglobin A1c (HbA1c) at 12 weeks | 12 weeks
  Hemoglobin A1c (HbA1c) measurements are calculated through fasting phlebotomy.
Change from baseline Plasminogen Activator Inhibitor-1 at 12 weeks | 12 weeks
  Plasminogen activator inhibitor type 1 (PAI-1) measurements are calculated through fasting phlebotomy.
Change from baseline Fibrinogen Antigen at 12 weeks | 12 weeks
  Fibrinogen Antigen measurements are calculated through fasting phlebotomy. High values indicate inflammation and increased risk of atherosclerosis.
Change from baseline Glucose at 12 weeks | 12 weeks
  Blood glucose measurements are calculated through fasting phlebotomy
Change from baseline high sensitivity C-Reactive Protein (hs-CRP) at 12 weeks | 12 weeks
  C-reactive protein measurements are calculated from blood samples collected through fasting phlebotomy.
Change from baseline Interleukin-6 (IL-6) at 12 weeks | 12 weeks
  IL-6 is calculated from blood samples collected through fasting phlebotomy
Change from baseline Creatinine at 12 weeks | 12 weeks
  Creatinine is calculated from blood samples collected through fasting phlebotomy
Change from baseline Cystanin C with eGFR at 12 weeks | 12 weeks
  Cystanin C with eGFR is calculated from blood samples collected through fasting phlebotomy
Change from baseline lipid panel at 12 weeks | 12 weeks
  Lipid panel measurements are calculated from blood samples collected through fasting phlebotomy.
Change from baseline 24-hour mean diastolic blood pressure at 12 weeks | 12 weeks
  Mean diastolic blood pressure over a 24-hour period is measured using an ambulatory blood pressure monitor.
Change from baseline 24-hour mean blood pressure at 12 weeks | 12 weeks
  Mean arterial blood pressure over a 24-hour period is measured using an ambulatory blood pressure monitor.
Change from baseline nocturnal mean systolic blood pressure at 12 weeks | 12 weeks
  Mean systolic blood pressure during sleep is measured using an ambulatory blood pressure monitor.
Change from baseline nocturnal mean diastolic blood pressure at 12 weeks | 12 weeks
  Mean diastolic blood pressure during sleep is measured using an ambulatory blood pressure monitor.
Change from baseline nocturnal mean blood pressure at 12 weeks | 12 weeks
  Mean arterial blood pressure during sleep is measured using an ambulatory blood pressure monitor.
Change from baseline Psychomotor Vigilance Task reaction time at 12 weeks | 12 weeks
  3-minute Psychomotor Vigilance Tasks will be done to quantify the speed with which subjects respond to a visual stimulus.
Change from baseline Psychomotor Vigilance Task lapses per test at 12 weeks | 12 weeks
  3-minute Psychomotor Vigilance Tasks will be done to quantify the speed with which subjects respond to a visual stimulus.
Change from baseline Functional Outcome of Sleep Questionnaire (FOSQ) at 12 weeks | 12 weeks
  This test will be used to assess the impact of excessive sleepiness on functional outcomes relevant to daily behaviors and sleep-related quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Ali Azarbarzin, PhD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol